CLINICAL TRIAL: NCT04174053
Title: Concordance Between Body Temperature Measured Per Enteric Capsule and Auricular Temperature in Neutropenic Patients Hospitalized in Intensive Hematology Care Units
Brief Title: Concordance Between 2 Means of Temperature Measure in Neutropenic Patients Hospitalized in Intensive Hematology Care Units
Acronym: TEMPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB18.09
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Haematological Malignancy
Keywords: Temperature measurement; capsule thermometers; Haematology
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temperature measurement (Experimental): enteric capsule will be ingested every 24 hours during aplasia. Temperature measurement will be made continuously during aplasia.
  In parallel, auricular temperature will be measure every 4 hours during aplasia.
  Interventions: Device: Enteric capsule

INTERVENTIONS:
Device: Enteric capsule — Enteric capsule to measure body temperature will be ingested every 24 hours during aplasia. the temperature measured with this technique will be compared with auricular temperature measurement (in current practice nurse measure temperature every 4 hours during aplasia).

SUMMARY:
Connected medicine "2.0" is a major challenge that will lead in the near future to profound changes in medical practices. Our study is part of this technological transformation, which is already taking the form of multiple devices available to practitioners: connected pill dispensers, integrated monitoring and surveillance systems (telemedicine), connected sensors, etc.

However, a symptom as crucial and simple as body temperature has not been measured by real-time enteric capsule in a context of neutropenia. We therefore wish to study the concordance between the peripheral (tympanic) temperature and that measured by a capsule ingested in a cohort of patients hospitalized in the USIH. If the measurements are clinically reliable and truly allow anticipation of antimicrobial treatments, a medico-economic evaluation will be proposed between the two options in the context of USIH before its possible generalization.

ELIGIBILITY:
Inclusion Criteria:

* Major patient admitted to USIH for an aplasia episode of at least 7 days secondary to:
* autograft conditioned by melphalan (MLP) or BEAM (BICNU, Etoposide, Aracytine, Melphalan) chemotherapy
* Aracytin chemotherapy High dose (HD) or intermediate dose (DI)
* Signed informed consent;
* Affiliated or beneficiary of a social protection scheme.

Exclusion Criteria:

* Diarrhea (> 3 stools /day) at the time of inclusion
* Occlusive syndrome at the time of inclusion or patient at risk of developing occlusive syndrome
* Persons with or likely to have intestinal disorders that may lead to obstruction of the digestive tract, including diverticulitis
* People with digestive tract motility disorders
* Persons equipped with a pacemaker or an electro-medical implant
* Weight < 40 kg or BMI > 30
* Patient for whom an MRI examination may be indicated during the trial period
* Patient with proven swallowing disorders
* Refusal to participate in the study
* Induction of acute leukaemia or allograft
* Person under guardianship or curatorship, or deprived of liberty by a judicial or administrative decision
* Pregnant, parturient or breastfeeding women;
* Patient unable to understand the study for any reason or to comply with the constraints of the trial (language, psychological, geographical problem, etc.)
* Patient who has already been included in the TEMPET trial during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the concordance between the body temperature measured at the periphery by ear thermometer and the body temperature measured per enteric capsule | 6 months
  the temperature in degrees Celsius measured by the 2 systems (left and right average for the auricular measure) and analysis of the concordance

SECONDARY OUTCOMES:
Estimate of the theoretical administration date of the anti-infective if enteral temperature had been taken into consideration | 6 months
  The time required to start anti-infective treatments according to the 2 measurement methods, in hours (effective start up thanks to the ear and theoretical measurement indicated by the enteric measurement)
Description of curves of temperature in the neutropenic patient measured continuously | 6 months
  Description of curves of temperature in the neutropenic patient measured continuously
Satisfaction of patient towards enteric capsule | 6 months
  auto-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, Professor, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No